CLINICAL TRIAL: NCT01037556
Title: Phase I/II Study of PR104 in Subjects With Refractory/Relapsed Acute Leukemia Using Adaptive Dose Selection
Brief Title: PR104 in Treating Patients With Refractory/Relapsed Acute Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Proacta, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR104-2004
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia
Keywords: AML; Acute Myeloid Leukemia; Acute Myelogenous Leukemia; Refractory AML; Relapsed AML; Refractory Acute Myeloid Leukemia; Relapsed Acute Myeloid Leukemia; Refractory Acute Myelogenous Leukemia; Relapsed Acute Myelogenous Leukemia; ALL; Acute Lymphocytic Leukemia; Relapsed Acute Lymphocytic Leukemia; Refractory Acute Lymphocytic Leukemia; Relapsed ALL; Refractory ALL
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: PR104 (Experimental)
  Interventions: Drug: PR104

INTERVENTIONS:
Drug: PR104 — Nine pre-defined dose levels for specific subsets of subjects will be administered by IV (in the vein). PR104 will be administered initially as induction therapy followed by administration as consolidation therapy, as is typical of established treatment regimens in AML.

SUMMARY:
The current understanding of PR104 justifies the evaluation of PR104 in subjects with relapsed/refractory AML and ALL. These include:

* Hypoxia. Leukemic bone marrow is likely to demonstrate a level of hypoxia sufficient to activate PR104 to its active metabolites PR104H and PR104M.
* Myelotoxicity as the primary toxicity at MTD. In prior clinical studies in subjects with solid tumors PR104 has demonstrated myelotoxicity as the primary toxicity. This observation suggests that PR104 will exert a similar effect on leukemic cells.
* AKR1C3. AML has been reported to exhibit high levels of AKR1C3 which should lead to selective activation of PR104 within both hypoxic and oxic leukemic cells.
* Preclinical data. PR104 has demonstrated impressive activity in an initial study using primary human ALL in a mouse model.

The initial dose finding phase of the study will provide estimates of the activity and toxicity of PR104 in subjects with refractory/relapsed AML, and determine the optimal individualized dose to give each subject based on his/her covariates (prior CR duration, prior number of salvage therapies, age). Once a potentially beneficial dose has been determined, an expanded cohort of subjects with AML or ALL will receive PR104 at a uniform dose. This information will prove valuable in defining the future clinical development of PR104, and in determining if PR104 has sufficient activity and acceptable safety in AML to warrant future phase II or phase III studies in this indication.

Primary objectives

* Determine the toxicities and recommended dose of PR104 when administered IV to subjects with relapsed/refractory AML and ALL.

Secondary objectives

* Evaluate the pharmacokinetics (PK) of PR104 and a series of PR104 metabolites
* Evaluate any anti-tumor effects of PR104
* Evaluate the expression of AKR1C3 in bone marrow and leukemic cells
* Evaluate potential biomarkers of hypoxia

DETAILED DESCRIPTION:
A single arm study defining the recommended dose of PR104 for each subpopulation in this patient population.

Following informed consent, subjects will undergo baseline evaluation with a history, physical exams, blood work, and disease assessment. Subjects will be assigned a dose of PR104 based on a Bayesian model maintained at the Statistical department at MD Anderson Cancer Center. The model will be updated with both toxicity and efficacy data as it is generated for each subject. New subjects will receive the currently predicted best dose for their respective subset based on prior treatment, age and duration of prior response.

PR104 will be administered initially as induction therapy for up to 3 cycles. Response will be assessed around day 42 (+/- 2 days) of the study. Subjects who obtain a CR or CRp will receive consolidation therapy for up to 4 additional cycles.

Subjects will be evaluated each week during the induction phase of the study. During the consolidation phase of the study, subjects will be evaluated on Day 1 of each cycle and as clinically indicated. Subjects with clinically significant progression will be removed from study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 18 years or more
* Histologically diagnosed acute myeloid leukemia (AML) or acute lymphocytic leukemia (ALL) by WHO classification
* Refractory or relapsed disease (requiring at least 5% leukemic blasts in the bone marrow, regardless of the presence of other features such as new or recurrent dysplastic changes or extramedullary disease) according to the following definitions:

AML Relapsed (defined as ≥5% leukemic blasts in the bone marrow) after receiving up to 2 prior induction regimens, (i.e., first or second relapse); Refractory (defined as ≥5% leukemic blasts in the bone marrow) to not more than 1 prior induction regimen (defined as failure to achieve a CR or CRp following induction therapy), (i.e., up to 1 induction failure).

ALL Relapsed/refractory (defined as ≥5% leukemic blasts in the bone marrow) after receiving 1 or more prior induction regimens, (i.e., any number of relapses)

* ECOG performance status of 0-2
* At least 2 weeks from administration of prior anti-leukemia therapy unless subject has progressed while receiving targeted therapy on a continuous dosing schedule
* No remaining clinically significant toxicities from prior chemotherapy of grade 2 or greater
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must be willing to use an acceptable contraceptive method (abstinence, oral contraceptive or double barrier device) for the duration of the study and for 30 days following the last dose of study drug, and must have a negative urine or serum pregnancy test within 2 weeks prior to beginning treatment on this trial
* Sexually active men must be willing to use an acceptable contraceptive method for the duration of time on study and for 30 days following the last dose of study drug
* Clinical laboratory values within the following ranges unless considered due to leukemic organ involvement: Serum creatinine 2.0 mg/dl; Total bilirubin 1.5x the upper limit of normal unless considered due to Gilbert's syndrome; Alanine aminotransferase (ALT), or aspartate aminotransferase (AST) 3x the upper limit of normal
* Willingness to provide at least one pre-PR104 leukemia sample (e.g., bone marrow or peripheral blood) for analysis of AKR1C3.

Exclusion Criteria:

* Pregnant and nursing subjects
* Uncontrolled intercurrent illness including, but not limited to uncontrolled infection, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Active heart disease including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, or uncontrolled congestive heart failure
* Another active concomitant malignancy likely to effect any of the primary or secondary outcome measures in the current study
* Subjects receiving any other standard or investigational treatment for their hematologic malignancy (other than hydroxyurea). Subjects with CNS leukemia are eligible and may receive concurrent standard intrathecal chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Determine the optimal individualized dose to give each refractory/relapsed AML subject based on his/her covariates (prior CR duration, prior number of salvage therapies, age). | 42 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Konopleva M, Thall PF, Yi CA, Borthakur G, Coveler A, Bueso-Ramos C, Benito J, Konoplev S, Gu Y, Ravandi F, Jabbour E, Faderl S, Thomas D, Cortes J, Kadia T, Kornblau S, Daver N, Pemmaraju N, Nguyen HQ, Feliu J, Lu H, Wei C, Wilson WR, Melink TJ, Gutheil JC, Andreeff M, Estey EH, Kantarjian H. Phase I/II study of the hypoxia-activated prodrug PR104 in refractory/relapsed acute myeloid leukemia and acute lymphoblastic leukemia. Haematologica. 2015 Jul;100(7):927-34. doi: 10.3324/haematol.2014.118455. Epub 2015 Feb 14. PMID 25682597